CLINICAL TRIAL: NCT03926520
Title: Effect and Safety of Electroconvulsive Therapy Plus Usual Care for the Acute Management of Severe Agitation in Dementia
Brief Title: Electroconvulsive Therapy (ECT) for Agitation in Dementia (AD)
Acronym: ECT-AD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brent Forester (Other)
Collaborators: Mayo Clinic (Other); Pine Rest Christian Mental Health Services (Other); Emory University (Other); The Zucker Hillside Hospital (Other); Medical University of South Carolina (Other)
Responsible Party: Sponsor-Investigator, Brent Forester, Principal Investigator, Mclean Hospital
Organization: Mclean Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020P002276
Record Dates: First submitted 2019-04-19; First posted 2019-04-24 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Alzheimer Dementia; Agitation,Psychomotor
Keywords: ECT; Agitation; Alzheimer's; Dementia
MeSH Terms: conditions — Alzheimer Disease; Psychomotor Agitation; Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- ECT+UC group (Experimental): ECT with Usual Care
  Interventions: Device: Electroconvulsive Therapy (ECT)

INTERVENTIONS:
Device: Electroconvulsive Therapy (ECT) — Stimulus method of delivery will be RUL electrode placement, and ultra-brief (UB) pulse width (0.25-0.37ms). At the first ECT session, seizure threshold (ST) will be determined by titration with the empirical dose titration method and subsequent treatments will be approximately 6 times the ST. Following other NIMH sponsored multicenter ECT studies (PRIDE, U01 MH055495), stimulus settings will be adjusted as needed during the ECT course based on seizure quality and treatment efficacy. Participants will be administered anesthesia.

SUMMARY:
This study will explore the effect of ECT treatments plus usual care (ECT+UC) in reducing severe agitation in patients with moderate to severe dementia including Alzheimer's Disease, Vascular dementia, Frontotemporal dementia, and Dementia with Lewy Bodies. The study will also determine the tolerability/safety outcomes of ECT+UC.

DETAILED DESCRIPTION:
This study will be a single-arm, unblinded, non-randomized trial to determine the effect and safety of ECT for severe agitation in moderate to severe stage dementia, while also examining the durability of the acute treatment effect in an exploratory maintenance naturalistic design. We plan to enroll 50 participants with an estimated dropout rate of 20%. We expect 50 participants to complete at least 1 ECT treatment before moving into the 12-month naturalistic follow-up phase.

ELIGIBILITY:
Inclusion Criteria

1. Diagnosis of Dementia, of the following subtypes,

   1. Alzheimer's dementia, according to NIA-AA Criteria for dementia
   2. Vascular dementia based on:

   i. History consistent with insidious onset of illness and gradual clinical decline ii. MRI evidence of microvascular ischemic disease (microinfarcts) iii. Physical and neurological examination do not indicate current or prior stroke c. Frontotemporal dementia d. Dementia with Lewy Bodies
2. Mini Mental Status Exam (MMSE) less than or equal to 15
3. Cohen-Mansfield Agitation Inventory Nursing Home Version (CMAI) score of 5 or more on at least one item or score of 4 on two items of aggression or physical nonaggression that holds potentially dangerous consequences including hitting (including self), kicking, grabbing onto people, pushing, throwing things, biting, scratching, spitting, hurting self or other, tearing things or destroying property, making physical sexual advances, trying to get to a different place, or intentional falling (items 1-11, 14, 15) OR one score of 5 or more in items of verbal aggression including screaming, making verbal sexual advances, and cursing or verbal aggression (items 22-24).
4. At least one failed pharmacological intervention to manage behavioral symptoms
5. Medically stable for safe administration of ECT verified by standard physical examination, urinalysis and serum chemistries and brain imaging when clinically indicated
6. Comprehension of English language
7. Authorized legal representative able and willing to give informed consent
8. Age 40 and above

Exclusion Criteria:

1. Current diagnosis of co-morbid delirium, measured by the Confusion Assessment Measure (CAM) and by clinical diagnosis
2. Diagnosis of vascular dementia due to stroke, based on:

   * History consistent with abrupt onset and step-wise progression of cognitive and functional decline
   * MRI scan within the past 12 months demonstrating evidence of hemorrhagic and embolic stroke
   * Physical and neurologic examination consistent with current or prior stroke
3. Lifetime or current diagnosis of Schizophrenia, Bipolar Disorder or Schizoaffective Disorder
4. Active substance use disorder within past 6 months
5. Treatment with ECT or other neurostimulation therapies (e.g., TMS or vagal nerve stimulation) within the past 3 months

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-01-28 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
CMAI total score | The CMAI will be collected through study completion, about 13 months
  The CMAI measures the efficacy of ECT+UC in reducing severe agitation in AD subjects. The CMAI is a 29-item scale with each item ranging from 1-7 in frequency with 7 being the highest and therefore worst outcome.

SECONDARY OUTCOMES:
Alzheimer's Disease Cooperative Study-Clinical Global Impression of Change Scale (ADCS-CGIC) | The ADCS-CGIC will be collected for one month
  The ADCS-CGIC gives a discrete score that ranges from 1-7 with 7 being the worst outcome.
Neuropsychiatric Inventory, Clinician Version (NPI-C) | The NPI-C will be collected for one month
  The NPI-C is an improved version of the NPI composed of several domains of which we will use Agitation and Aggression, as well as their sum. The higher the frequency and/or severity within each domain, the worse the condition of the patient.
Pittsburgh Agitation Scale (PAS) | The PAS will be collected for one month
  The PAS assesses four behavioral domains. Each domain has an intensity score ranging from 0-4 with 4 being the worst outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Brent P Forester, MD, MSc, Principal Investigator — Mclean Hospital; George Petrides, MD, Principal Investigator — Northwell Health
Locations (5):
- United States (5):
  - Emory Healthcare, Atlanta, Georgia
  - McLean Hospital, Belmont, Massachusetts
  - Pine Rest Christian Mental Health Services, Grand Rapids, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Northwell Health, Glen Oaks, New York